CLINICAL TRIAL: NCT07350460
Title: A Randomized, Double-Blind Trial Comparing Pudendal Block Versus Sacral ESP for Ambulatory Hemorrhoidectomy
Brief Title: PUSHES (Pudendal Block Versus Sacral ESP Hemorrhoidectomy Study)
Acronym: PUSHES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Saporito (Other)
Responsible Party: Sponsor-Investigator, Andrea Saporito, Prof. Dr. Med., Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PUSHES trial
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Hemorrhoids; Hemorrhoids Third Degree
Keywords: Hemorrhoids; Hemorrhoidectomy; Postoperative Pain; Pain Measurement
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pudendal block (Active Comparator): Patients in the control group will receive an ultrasound-guided bilateral pudendal nerve block with 20 mL of 0.75% ropivacaine and a sacral ESP block with 20 mL of normal saline. Blinding is ensured by the double block procedure
  Interventions: Procedure: Pudendal block AL; Procedure: Sacral ESP block Sham
- Sacral ESP block (Experimental): Patients in the intervention group will receive an ultrasound-guided sacral ESP block with 20 mL of 0.75% ropivacaine and a bilateral pudendal nerve block with 20 mL of normal saline.
  Interventions: Procedure: Sacral ESP block AL; Procedure: Pudendal block Sham

INTERVENTIONS:
Procedure: Pudendal block AL — Patients in the control group will receive an ultrasound-guided bilateral pudendal nerve block with 20 mL of 0.75% ropivacaine
  Arms: Pudendal block
Procedure: Sacral ESP block AL — Patients in the intervention group will receive an ultrasound-guided sacral ESP block with 20 mL of 0.75% ropivacaine
  Arms: Sacral ESP block
Procedure: Sacral ESP block Sham — Patients in the control group will receive a sacral ESP block with 20 mL of normal saline.
  Arms: Pudendal block
Procedure: Pudendal block Sham — Patients will receive a bilateral pudendal nerve block with 20 mL of normal saline.
  Arms: Sacral ESP block

SUMMARY:
The goal of this clinical trial is to learn if the sacral erector spinae plane block can provide equal or better pain control than the pudendal nerve block in adults undergoing hemorrhoid surgery. The main question is: Which block offers more effective analgesia and faster recovery?

DETAILED DESCRIPTION:
Hemorrhoidectomy remains one of the most common anorectal procedures performed worldwide, yet it is frequently associated with significant postoperative pain that can impair recovery, delay discharge, and increase unplanned healthcare utilization. Effective analgesia is therefore a central component of perioperative care in this population.

Traditionally, the pudendal nerve block has been used to provide postoperative analgesia after hemorrhoidectomy. While effective, this technique requires precise anatomical identification, can be technically challenging, and is associated with potential risks such as vascular puncture or local anesthetic systemic toxicity. More recently, the sacral erector spinae plane (ESP) block has been described as a simpler, ultrasound-guided technique that may provide effective analgesia for procedures involving the perineal and anorectal region. Its safety profile and ease of performance could represent an attractive alternative to the pudendal nerve block, especially in the ambulatory setting.

The PUSHES trial is designed as a randomized, controlled, double-blind study to directly compare the efficacy of sacral ESP block versus pudendal nerve block for pain control after ambulatory hemorrhoidectomy. A total of 64 adult patients undergoing elective hemorrhoidectomy under standardized spinal anesthesia will be enrolled. Following spinal anesthesia, participants will be randomized to receive either a sacral ESP block with ropivacaine and a sham pudendal block with saline, or a pudendal block with ropivacaine and a sham sacral ESP block with saline. This double-dummy design ensures blinding of patients, anesthesiologists, and outcome assessors.

The primary endpoint is pain intensity at 4 hours postoperatively, measured using a 10-point Visual Analog Scale (VAS). Secondary endpoints include pain scores at 12 and 24 hours, time to first rescue analgesia, opioid consumption, functional recovery milestones (mobilization, ability to void, return to baseline activity), and block-related or systemic adverse events.

By systematically comparing these two techniques, this trial aims to identify whether the sacral ESP block can provide equivalent or superior analgesia to the pudendal nerve block while offering a simpler, safer alternative for routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) scheduled for elective excisional hemorrhoidectomy;
* Ability to understand the nature of the study and provide written informed consent;
* American Society of Anesthesiologists (ASA) physical status I-III;
* Ability to comply with study procedures and postoperative evaluations.

Exclusion Criteria:

* Pregnancy;
* Body weight under 50 kg due to the potential risk of local anaesthetic systemic toxicity (LAST);
* BMI > 40; Known allergy or contraindication to local anaesthetics (e.g., ropivacaine, prilocaine);
* Severe coagulation disorders or current anticoagulant therapy contraindicating spinal or peripheral deep nerve blocks (like pudendal block, because Sacral ESP is considered a superficial block);
* Infection at the puncture site;
* Neurological disorders affecting the sacral or pudendal nerve pathways;
* Severe psychiatric conditions impairing study participation;
* Language barriers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2027-09-29 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity, assessed using the Visual Analogue Scale (VAS) at 4 hours following surgery in day 0 | Day 0

SECONDARY OUTCOMES:
VAS (Visual Analogue Score) pain scores at 12 hours and 24 hours postoperatively | Day 0 and day 1
Time to first request for rescue analgesia in 24 hours | Day 0 and day 1
Total amount of rescue analgesia in 24 hours | Day 0 and day 1

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Saporito, Prof. Dr. Med., Study Chair — Department of Anesthesiology, Ospedale San Giovanni, Ente Ospedaliero Cantonale, Bellinzona, Switzerland
Locations (1):
- Ospedale Regionale Bellinzona e Valli (ORBV) CH-6500 Bellinzona Switzerland, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared upon reasonable request from qualified investigators by contacting the Principal Investigator via email. Due to the double-blind design of the study, raw data will not be shared before study completion, unblinding, and final statistical analyses. Following these steps, de-identified individual-level data may be made available to support requests aimed at verifying or challenging the reported findings, subject to appropriate scientific justification and compliance with applicable data protection regulations.

REFERENCES:
- [Result] Kaya C, Dost B, Tulgar S. Sacral Erector Spinae Plane Block Provides Surgical Anesthesia in Ambulatory Anorectal Surgery: Two Case Reports. Cureus. 2021 Jan 9;13(1):e12598. doi: 10.7759/cureus.12598. PMID 33585088